CLINICAL TRIAL: NCT05998057
Title: The Effect of Neuromuscular Exercise Training on Balance, Jump and Trunk Endurance in Female Ice Hockey Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar70
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Sports Physical Therapy
Keywords: Ice hockey; Neuromuscular exercise; Vertical jump; Trunk endurance; Y balance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The intervention group will be given neuromuscular exercises 5 days a week for 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: The control group will be asked to continue the standard (routine) classical training training (5 days/12 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The control group was asked to continue the standard (routine) classical training training (5 days/12 weeks).
  Interventions: Other: control
- exercise group (Experimental): The neuromuscular training program has been adapted to ice hockey players. The content of the program includes core stabilization, balance and plyometric exercises. The session duration was set to be approximately 60-90 minutes. An average session is 15 minutes of warm-up, followed by 30-40 minutes. continued with neuromuscular training program, 15 min. It was ended with cooling and stretching exercises. Since all exercises are done with body weight, no extra equipment is needed.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Exercises:
  Lunge to Hamstrings Stretch 3 sets of 30 seconds
  * Standing Hip Out 3 sets of 30sec
  * 90-90 Hip Stretch 3 sets of 30 seconds
  * World's Greatest Stretch 3 sets of 30 seconds
  * Star Excursion 3 sets of 5 reps
  * Side Jumps+ Balance 3 sets of 10 reps
  * Forward Hops + Balance 3 sets of 10 reps
  * Squat 3 sets of 10 reps
  * Squat Jump 3 sets of 10 reps
  * Jumping Spider Push-up 3 sets of 10 reps
  * Double Leg Vertical Jump 3 sets of 10 reps
  * Broad Jumps 3 sets of 10 reps
  * Lateral Box Shuffles 3 sets of 10 reps
  * Plank 3 sets of 30 seconds
  * Side Plank 3 sets of 30 seconds
  * Bird Dog 3 sets of 10 reps
  * Glute Bridge 3 sets of 10 reps
  * Single Leg Glute Bridge 3 sets of 10 reps
  * Single Toe Raises 3 sets of 30sec
  * Nordic Hamstrings 3 sets of 10 reps
  * Monster Walk 3 sets of 10 reps
  Arms: exercise group
Other: control — The control group was asked to continue the standard (routine) classical training training (5 days/12 weeks).
  Arms: control group

SUMMARY:
The aim of the study is to investigate the changes in dynamic balance, vertical jump and trunk endurance parameters in athletes included in body weight neuromuscular program in addition to regular training programs.

DETAILED DESCRIPTION:
As a randomization method, the participants will be divided into two groups as control and experimental groups by using a computer-based program and a simple randomization method. This study will be scheduled five times a week for six weeks. After the evaluations, all exercises will be taught to the experimental group by the physiotherapist. While the experimental group will apply to this program and traditional education, the control group will continue to the traditional education program. Since all exercises are done with body weight, no extra equipment will be needed. Reviews:

Balance evaluation: Y balance test The Vertical Jump Test will be used to evaluate muscle strength in the lower extremities.

McGill Trunk Endurance Test: To be used for Muscular Endurance Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed athlete of any team affiliated with the Turkish Ice Hockey Federation and competing in the league,
* Athletes who do not use any medication and do not have a medical condition that would interfere with the tests
* be between the ages of 15-30

Exclusion Criteria:

* Not having had a musculoskeletal injury in the last 1 year that would prevent him from training or that would affect the results of the measurements.

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Y balance test | 13 weeks
  The test is a practical functional test that can predict dynamic balance and postural stability. The player's performance improves with balance, flexibility, coordination and power integration. For this test, players stand in the center of a 'Y' shaped arrangement with 3 lines drawn at certain angles. The players are asked to reach in anterior, posterolateral and posteromedial directions using one foot. Three applications are made in each direction and the average of the reach distances is recorded in centimeters. Pre-measured leg length is used to normalize the mean score of these three treatments. Percentage of maximum reach = deflection distance/leg length. Leg length; Spina iliaca anterior superior to the distal point of the medial malleolus. To obtain an overall measure of the Y Balance Test, data from all directions must be averaged to calculate the composite score.
Vertical Jump Test | 13 weeks
  The Vertical Jump Test is used to evaluate muscle strength in the lower extremities. The maximum jump height reached gives information about the muscle strength and functional capacity of the lower extremities in many sports. The player keeps the feet flat on the ground. The point of the fingertips reached is recorded. This is called standing reach height. The player then begins in a stance with the knees extended, standing away from the wall, feet shoulder-width apart. After the player flexes their knees and hips, they jump up and reach the highest point they can reach with their hands. The test is performed three times and the highest distance is used as the jump height.
McGill Body Endurance Test | 13 weeks
  For trunk flexors, extensors and lateral muscles, a series of isometric tests showing the endurance of trunk muscles have been defined. The test consists of 3 parts. There is a 5-minute break between each test.
  Tests:
  * Trunk Flexor Muscle Endurance Assessment
  * Right and Left Lateral Trunk Muscle Endurance Assessment
  * Back Extensor Muscle Endurance Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Merve KAPANŞAHİN, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ransdell LB, Murray T. A physical profile of elite female ice hockey players from the USA. J Strength Cond Res. 2011 Sep;25(9):2358-63. doi: 10.1519/JSC.0b013e31822a5440. PMID 21804420
- [Background] Ronnestad BR, Ofsteng SJ, Ellefsen S. Block periodization of strength and endurance training is superior to traditional periodization in ice hockey players. Scand J Med Sci Sports. 2019 Feb;29(2):180-188. doi: 10.1111/sms.13326. Epub 2018 Nov 8. PMID 30350896
- [Background] Roczniok R, Stanula A, Maszczyk A, Mostowik A, Kowalczyk M, Fidos-Czuba O, Zajac A. Physiological, physical and on-ice performance criteria for selection of elite ice hockey teams. Biol Sport. 2016 Mar;33(1):43-8. doi: 10.5604/20831862.1180175. Epub 2015 Nov 19. PMID 26985133
- [Background] Burr JF, Jamnik RK, Baker J, Macpherson A, Gledhill N, McGuire EJ. Relationship of physical fitness test results and hockey playing potential in elite-level ice hockey players. J Strength Cond Res. 2008 Sep;22(5):1535-43. doi: 10.1519/JSC.0b013e318181ac20. PMID 18714234
- [Background] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287